CLINICAL TRIAL: NCT01905735
Title: A Multicentric,Double-blind,Placebo Controlled,Phase-2 Study to Assess the Safety and Efficacy of Homeopathic Medicine Rhus Toxicodendron 30 in the Treatment of Rheumatoid Arthritis .
Brief Title: A Safety and Efficacy of Homeopathic Medicine Rhus Toxicodendron 30 in the Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthcare Homoeo Charitable Society (Other)
Responsible Party: Principal Investigator, ravinder kochhar, principal investigator, Healthcare Homoeo Charitable Society
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLSGB-01
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis.
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): 1/2 ml of dispensing alcohol administered orally at every 7 day for 5 month .
  Interventions: Drug: placebo
- Rhustoxicodendron 30 (Active Comparator): 1/2ml Rhustoxicodendron 30 is administered orally every 7 day for 5 month.
  Interventions: Drug: Rhustoxicodendron 30

INTERVENTIONS:
Drug: Rhustoxicodendron 30 — 1/2ml Rhustoxicodendron 30 is administered orally every 7 day for 5 month.
  Other Names: poison ivy
  Arms: Rhustoxicodendron 30
Drug: placebo — 1/2 ml of dispensing alcohol is administered every 7 day for 5 month orally.
  Other Names: dispensing alcohol
  Arms: placebo

SUMMARY:
the purpose of the study is to assess the safety and efficacy of commonly used Homeopathic medicine Rhustoxicodendron in 30 potency in the treatment of Rheumatoid arthritis.

DETAILED DESCRIPTION:
it is a multicenter phase 2 ,double blind study in patient with active Rheumatoid arthritis ,there are 2 group in the study A and B ,where group A receive Rhustoxicodendron in 30 potency the first dose will administered orally (1/2 ml)after the completion of case taking ,and repeated every 7th day for 5 month and on the other hand group B receive placebo orally in (1/2 ml) at same interval for same period .

ELIGIBILITY:
Inclusion Criteria:

* those who will provide written consent to participate in the study
* patient willing to turn up for 7th day follow up
* patient who are willing and compliance to the study
* those who are between 25 to 60 years .
* patient who are willing and compliance to the study .
* ESR more then 28 mm.

Exclusion Criteria:

* Participating as a subject in any other clinical research study.
* Children below the age of 25years.
* Female subject who are pregnant or planning for pregnancy within 6 month.
* History of seizures
* Breast feeding women's.
* Patient on treatment for life threatening illness like cancer aids etc.
* Patient should not have any congenital abnormality or patient should not have undergone any operative procedure as consequences of RA.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Number of subject With American College of Rheumatology (ACR) Criteria Improvement of at Least 20%, 50%, and 70% (ACR 20/50/70 Responders). | 6 weeks upto 24 week
  number of subject with ACR criteria improvement consisting of ACR 20,ACR50,ACR70 reduction in tender and swollen joint counts and 20%,50%,70% improvement respectively in 3 of the following 5 criteria .
  1. physician global assessment of disease activity's.
  2. patient global assessment of disease activity's.
  3. subject assessment of pain
  4. subject assessment of function disability via health assessment questionnaire[HAQ]
  5. acute phase reactant ESR every 6 weeks upto 24 week

SECONDARY OUTCOMES:
mean change from baseline in tender joint count. | 6 weeks upto 24 week
mean change from baseline in swollen joint. | 6 weeks upto 24 week
mean change from baseline in physician global assessment of disease activity. | every 6 weeks upto 24 week
  mean change from baseline in physician assessment of disease activity via visual analog scale(0-100 mm)
mean change from baseline in patient global assessment of disease . | 6 weeks upto 24 week
  mean change from baseline in patient global assessment of disease via visual analog scale(0-100 mm)
mean change from baseline in subject assessment of pain using VAS from 0-100 mm | 6 weeks upto 24 week
mean change from baseline in ESR | 6 weeks upto 24 week
mean change from baseline in disability index of the health assessment Questionnaire (HAQ) | 6 weeks upto 24 week

CONTACTS AND LOCATIONS:
Overall Officials: ravinder kochhar, MD hom, Principal Investigator — Healthcare Homoeo Charitable Society; mukesh k singh, B.H.M.S, Study Director — health care homoeo charitable society
Locations (2):
- India (2):
  - Gupta Homoeo Clinic, Delhi, National Capital Territory of Delhi
  - Kochhar Clinic, Ludhiana, Punjab